CLINICAL TRIAL: NCT02920684
Title: Haemodynamic and Metabolism Response During Early Rehabilitation in Sedated Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Principal Investigator, BOUCHRA LAMIA, MD, PhD, University Hospital, Rouen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-A01633-46
Record Dates: First submitted 2016-09-25; First posted 2016-09-30 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Critically Ill Patients Under Mechanical Ventilation; Sedated Patients
Keywords: Early rehabilitation; Mechanical ventilation; Physiotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Passive legs mobilisation (Active Comparator): A physiotherapist performs passive legs movement
  Interventions: Other: Passive legs mobilisation
- Passive cycloergometer (Active Comparator): A motorized cycloergometer performs passive legs cycling
  Interventions: Other: Passive cycloergometer
- Muscular electrical stimulation (Active Comparator): Quadriceps neuromuscular electrical stimulation
  Interventions: Other: Muscular electrical stimulation
- FES cycling (Active Comparator): A motorised cycloergometer performs a quadriceps neuromuscular electrical stimulation during passive
  Interventions: Other: FES cycling

INTERVENTIONS:
Other: Passive legs mobilisation — A physiotherapist performs a passive leg movement
  Arms: Passive legs mobilisation
Other: Passive cycloergometer — A motorised cycloergometer performs a passive cycling
  Arms: Passive cycloergometer
Other: Muscular electrical stimulation — A neuromuscular electrical stimulation device performs a quadriceps located stimulation
  Arms: Muscular electrical stimulation
Other: FES cycling — A motorised cycloergometer performs a passive cycling with quadriceps neuromuscular stimulation
  Arms: FES cycling

SUMMARY:
Despite several positive studies, benefits of early rehabilitation on recovery and motor performance improvement need to be demonstrate. A recent study finds that despite early rehabilitation, 1 survivor of 2 (52%) acquired an ICU weakness. The low intensity exercises applied in intensive care is common and most patients stay in bed.

Under these conditions, the optimal choice of the rehabilitation technique for bedridden patient and its intensity should be studied.

The objective of the study is to evaluate the cardiovascular and metabolic response of patients during four interventions: Passive legs mobilization, Passive cycloergometter, Quadriceps neuromuscular electrical stimulation and Functional electrical stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation
* Sedated
* Ramsay < 4

Exclusion Criteria:

* Rehabilitation contraindication
* Patient with pacemaker
* Patient under volume assist control
* FiO2 > 80%
* Patient under neuromuscular blockers
* Neurologic comorbidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Cardiac output by cardiac ultrasonography | Every 3 minutes during 10 minutes exercise

SECONDARY OUTCOMES:
Muscular oxygenation of vastus lateralis muscle by Near Infrared Spectroscopy | Continuously during ten minutes exercise
Pulmonary artery Pressure by cardiac ultrasonography | Every 3 minutes during 10 minutes exercise
Tricuspid annular plane systolic excursion by cardiac ultrasonography | Every 3 minutes during 10 minutes exercise
Expiratory volume | Continuously during ten minutes exercise
Respiratory rate | Continuously during ten minutes exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Le Havre, Jacques Monod Hospital, Montivilliers, France

REFERENCES:
- [Derived] Medrinal C, Combret Y, Prieur G, Robledo Quesada A, Bonnevie T, Gravier FE, Dupuis Lozeron E, Frenoy E, Contal O, Lamia B. Comparison of exercise intensity during four early rehabilitation techniques in sedated and ventilated patients in ICU: a randomised cross-over trial. Crit Care. 2018 Apr 27;22(1):110. doi: 10.1186/s13054-018-2030-0. PMID 29703223
- [Derived] Medrinal C, Combret Y, Prieur G, Robledo Quesada A, Bonnevie T, Gravier FE, Frenoy E, Contal O, Lamia B. Effects of different early rehabilitation techniques on haemodynamic and metabolic parameters in sedated patients: protocol for a randomised, single-bind, cross-over trial. BMJ Open Respir Res. 2017 Jan 30;4(1):e000173. doi: 10.1136/bmjresp-2016-000173. eCollection 2017. PMID 28255448